CLINICAL TRIAL: NCT02226185
Title: A Randomized, Placebo-controlled, Multicenter, Prospective Clinical Study of Berberine Hydrochloride in Preventing Recurrence and Carcinogenesis After Endoscopic Removal of Colorectal Adenomas
Brief Title: Study of Berberine Hydrochloride in Prevention of Colorectal Adenomas Recurrence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jing-yuan Fang, MD, Ph. D, Director of Department of Gastroenterology, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RJ2014BH
Record Dates: First submitted 2014-08-23; First posted 2014-08-27 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Adenoma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Berberine hydrochloride (Experimental): supplement of Berberine hydrochloride 0.3g two times per day for 2-3 years
  Interventions: Drug: Berberine hydrochloride
- placebo (Placebo Comparator): identical-appearing placebo supplements for 2-3 years
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Berberine hydrochloride — supplement of Berberine hydrochloride 0.3g two times per day for 2-3 years
  Arms: Berberine hydrochloride
Drug: placebo — supplement of placebo two times per day for 2-3 years
  Arms: placebo

SUMMARY:
Berberine hydrochloride is a conventional component in Chinese medicine. In recent years, anticancer activity of berberine hydrochloride have been explored. The aim of this study is to investigate the effect of berberine hydrochloride on the recurrence of colorectal adenomas.

DETAILED DESCRIPTION:
Colorectal adenomas are well-known to be precancerous lesions that develop into colorectal cancers on the basis of the adenoma-carcinoma sequence. The effects of screening for colorectal adenomas and removing precancerous lesions on the prevention of colorectal cancer have been established. Because of the high recurrence rates of colorectal adenomas in patients who have undergone polypectomy, the potential chemopreventive agents that may reduce the risk of colorectal adenoma recurrence need to be investigated.

Berberine hydrochloride is a conventional component in Chinese medicine. In recent years, anticancer activity of berberine hydrochloride have been explored. The aim of this study is to investigate the effect of berberine hydrochloride on the recurrence of colorectal adenomas by conducting a randomized, placebo-controlled, prospective clinical.

ELIGIBILITY:
Inclusion criteria

* Individuals aged 18-75 years
* Individuals who had at least one and no more than 6 histologically confirmed CRAs removed within 6 months before recruitment
* Individuals who are able to swallow pills
* Individuals who voluntarily sign the consent form after being fully informed and understanding the purpose and procedure of this study, characters of the disease, effect of medication, methods of related examinations, and potential risk/benefits of the study 4.2 Exclusion criteria
* Individuals whose adenoma was not completely removed during previous colonoscopy
* Individuals with a history of familial adenomatous polyposis (FAP) or hereditary non-polyposis colorectal cancer (HNPCC, Lynch syndrome)
* Individuals who are taking regularly aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), cyclo-oxygenase 2 (COX2) inhibitors, calcium or vitamin D
* Individuals with a history of subtotal/total gastrectomy or partial bowel resection
* Individuals who are intolerant to another colonoscopy examination
* Individuals who are hypersensitive or intolerant to the drugs
* Individuals with severe heart, liver or kidney disease, or any cancer history
* Individuals presenting severe constipation
* Pregnant women, women during breast-feeding period, or women with expect pregnancy
* Individuals with mental diseases who are not able to cooperate
* Individuals who are involved in designing, planning or performing this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1108 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-12-29 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
Recurrence rates of CRA | until the last patient reached the 2 years follow-up
  The primary objective of this study is to investigate recurrence rates of colorectal adenoma (CRA) after Berberine hydrochloride or placebo intervention.

SECONDARY OUTCOMES:
The incidence of all polypoid lesions or advanced colorectal adenoma or colorectal cancer | until the last patient reached the 2 years follow-up
  The incidence of all polypoid lesions or advanced colorectal adenoma or colorectal cancer after Berberine hydrochloride or placebo intervention

OTHER OUTCOMES:
Changes in fecal microflora | baseline, the 1st year and the 2nd year
  Fecal microflora tests

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Yuan Fang, M.D., Ph.D, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (7):
- China (7):
  - Department of Gastroenterology, the Seventh Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Department of Gastroenterology, Zhongshan Hospital, Xiamen University, Xiamen, Fujian
  - Department of Gastroenterology, Nanfang Hospital, Southern Medical Univerisity, Guangdong, Guangzhou
  - Division of Gastroenterology and Hepatology, The Affiliated DrumTower of Nanjing University Medical School, Nanjing, Jiangsu
  - Division of Gastroenterology and Hepatology, Ren-Ji Hospital, Shanghai Jiao-Tong University School of Medicine, Shanghai Institute of Digestive Disease; Key Laboratory of Gastroenterology & Hepatology, Ministry of Health, Shanghai, Shanghai Municipality
  - Department of Gastroenterology, the Shanghai Tenth People's Hospital, Tongji University, Shanghai, Shanghai Municipality
  - Department of Gastroenterology and Hepatology, General Hospital, Tianjin Medical University, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Qian Y, Kang Z, Zhao L, Chen H, Zhou C, Gao Q, Wang Z, Liu Q, Cui Y, Li X, Chen Y, Zou T, Fang J. Berberine might block colorectal carcinogenesis by inhibiting the regulation of B-cell function by Veillonella parvula. Chin Med J (Engl). 2023 Nov 20;136(22):2722-2731. doi: 10.1097/CM9.0000000000002752. Epub 2023 Aug 9. PMID 37553874
- [Derived] Chen YX, Gao QY, Zou TH, Wang BM, Liu SD, Sheng JQ, Ren JL, Zou XP, Liu ZJ, Song YY, Xiao B, Sun XM, Dou XT, Cao HL, Yang XN, Li N, Kang Q, Zhu W, Xu HZ, Chen HM, Cao XC, Fang JY. Berberine versus placebo for the prevention of recurrence of colorectal adenoma: a multicentre, double-blinded, randomised controlled study. Lancet Gastroenterol Hepatol. 2020 Mar;5(3):267-275. doi: 10.1016/S2468-1253(19)30409-1. Epub 2020 Jan 8. PMID 31926918

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT02226185/Prot_SAP_001.pdf